CLINICAL TRIAL: NCT00114803
Title: Use of Intranasally Administered Calcitonin in the Treatment of Osteopenia and Osteoporosis in Children, Adolescents and Young Adults With IBD: A Pilot Study
Brief Title: Nasal Calcitonin in the Treatment of Bone Mineral Loss in Children and Adolescents With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Crohn's and Colitis Foundation (Other); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Calcitonin 1.0; CCFA #249
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-04

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: bone mineral density; osteoporosis; osteopenia; children; adolescents; DXA
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Osteoporosis; Bone Diseases, Metabolic

INTERVENTIONS:
Drug: Calcitonin nasal spray (salmon)

SUMMARY:
The hypothesis underlying this study is that nasally administered calcitonin will stabilize or improve bone mineral density in young patients with ulcerative colitis or Crohn's disease. Patients who participate will receive either calcitonin or placebo and will have their bone mineral density measured at the start, at nine months, and at 18 months of study. Participants will also receive age appropriate doses of vitamin D and calcium supplements. Other serological measures of vitamin D status will be obtained every 3 months during the study.

DETAILED DESCRIPTION:
This is an institutional, randomized, placebo-controlled, double-blind clinical trial to compare the efficacy of intranasally administered calcitonin (plus oral supplements of age-appropriate doses of calcium and vitamin D) with that of placebo nasal spray (plus oral supplements of age-appropriate doses of calcium and vitamin D) in maintaining or improving bone mineral density. Study subjects will be 8 to 22 year old patients with the diagnosis of inflammatory bowel disease (ulcerative colitis and Crohn's disease) and low bone mineral density defined as DXA z score lower than -1.0 SD. Study end-point will be at 18 months after the continuous administration of nasal calcitonin or placebo and supplements as above. Bone mineral density will be measured by dual energy X-Ray absorptiometry (DXA) at the beginning of the study, and then at 9 and 18 months. The study subjects will be evaluated clinically and nutritionally at the beginning of the study, as well as every 3 months for the duration of the study. Laboratory values relevant to calcium homeostasis and bone turnover will be obtained every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Low bone mineral density as defined
* Age 8 to 22 years
* Diagnosis of Crohn's disease or ulcerative colitis

Exclusion Criteria:

* Receiving calcitonin or biphosphonates, androgens or growth hormone
* Steroid induced fracture in the past
* Pregnant
* Diagnosis of kidney failure, polycystic ovaries syndrome, or malignancy

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66
Dates: Start 2004-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Bone mineral density at 18 months

SECONDARY OUTCOMES:
Bone mineral density at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States